CLINICAL TRIAL: NCT02444767
Title: A PK Study to Assess the Relative Systemic Exposure to Bimatoprost and Bimatoprost Acid After Administration of a Single 13 mg Bimatoprost Ocular Insert for 1 Week in Medically Stable Adult Subjects With or Without Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Bimatoprost Ocular Insert Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FSV5-006
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13mg Bimatoprost Insert (Experimental): Subjects in this arm have 13mg Bimatoprost Ocular Inserts placed in both eyes for 7 days.
  Interventions: Drug: 13mg Bimatoprost Ocular Insert

INTERVENTIONS:
Drug: 13mg Bimatoprost Ocular Insert — 13mg Bimatoprost Ocular Insert in each eye.

SUMMARY:
The Bimatoprost Ocular Insert is intended to provide sustained delivery of bimatoprost to the ocular surface to lower the intraocular pressure (IOP) in patients with open-angle glaucoma or ocular hypertension.

This study will evaluate the pharmacokinetic aspects of the Bimatoprost Ocular Insert in healthy (non-glaucoma) subjects.

DETAILED DESCRIPTION:
This study is designed to provide pharmacokinetic (PK) data with respect to the relative systemic exposure to bimatoprost and bimatoprost acid after administration of a single 13 mg Bimatoprost Ocular Insert for 1 week in medically stable adult subjects with or without primary open angle glaucoma (POAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 and 55 years, inclusive.
2. Subjects who are medically stable with or without POAG or OHT.
3. Written informed consent to participate in the study.
4. Body mass index between 18 and 30 kg/m², inclusive.
5. Female subjects of childbearing potential - not surgically sterile or at least 2 years postmenopausal - must agree to utilize one of the following forms of contraception from screening through completion of the study: abstinence, intrauterine device or vasectomized partner (6 months minimum).

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. A history of allergic or adverse responses to bimatoprost or any comparable or similar product.
3. Subjects who are unable to tolerate the Inserts that do not contain drug for the 7 days trial wear period.
4. Subjects who require two (2) or more site-assisted replacements of the inserts that do not contain drug during the 7 days trial wear period.
5. Subjects who will require contact lens use during the study period.
6. Subjects who currently have punctal occlusion in one or both eyes.
7. Subjects who have made a blood donation of one (1) pint or more within 30 days prior to study initiation.
8. Subjects who have made a plasma donation within 14 days of study initiation.
9. Participation in a clinical trial within 30 days prior to the first dose of Study Drug.
10. Use of any over-the-counter (OTC) medication, including vitamins, herbal products, and dietary supplements, during the study.
11. Use of any prescription medication during the medication washout (screening) period or during the study.
12. Required use during study of ocular medications or artificial tears.
13. Ocular, orbital, and/or eyelid surgery of any type within the past 6 months from screening date.
14. Past history of incisional surgery for glaucoma at any time.
15. Past history of corneal refractive surgery.
16. Any active ocular disease that in the opinion of the Investigator would interfere with the conduct of the study (e.g., severe dry eye, uveitis, inflammation, ocular infection, corneal edema). Patients may have mild blepharitis, mild dry eye, cataracts, age-related macular degeneration or background diabetic retinopathy if, in the opinion of the Investigator, it would not interfere with the conduct of the study.
17. Smoking or use of tobacco products or products containing nicotine within 6 months prior to or during the study.
18. Female subjects who are lactating.
19. Positive pregnancy test prior to administration of Study Insert for all women of childbearing potential.
20. Positive urine screen for alcohol, drugs of abuse, or cotinine.
21. Subjects with POAG or OHT for whom, in the opinion of the investigator, it would be unsafe to discontinue ocular hypotensive treatment for the required periods during the study.
22. Significant risk of angle closure due to pupil dilation, defined as a Shaffer classification of less than grade 2 based on gonioscopy performed within the last 12 months.
23. Subjects who were on ocular hypotensive treatment who are not fully washed out prior to receiving active inserts.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Whole blood concentrations of bimatoprost and bimatoprost acid | 7 days
  Whole blood concentrations of bimatoprost and bimatoprost acid will be measured using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Walker, PhD, Study Director — ForSight Vision 5
Locations (1):
- Sall Medical Research Center, Artesia, California, United States